CLINICAL TRIAL: NCT05459194
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, 3-way Crossover, Single Dose Study, Comparing the Efficacy and Safety of Fluticasone/Salmeterol Administered With Elpenhaler Versus Seretide Diskus in Patients With Asthma
Brief Title: Efficacy and Safety Study of Fluticasone/Salmeterol Administered With Elpenhaler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2007-FLUSAL-EL-01; 2008-000193-21 (EudraCT Number); Sponsor ID (Other: FLUSAL-01)
Record Dates: First submitted 2011-10-12; First posted 2022-07-14 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Asthma
Keywords: respiratory; combination treatment; Elpenhaler; Diskus
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Active Comparator): Fluticasone/Salmeterol Elpenhaler active vs Fluticasone/Salmeterol Diskus placebo
  Interventions: Device: RP - TA
- Refere (Placebo Comparator): Fluticasone/Salmeterol Elpenhaler placebo vs Fluticasone/Salmeterol Diskus active
  Interventions: Device: RP - TA

INTERVENTIONS:
Device: RP - TA — randomized, double-blind, double-dummy, placebo-controlled, 3-way crossover, single dose study, comparing the efficacy and safety of the Fluticasone/Salmeterol combination administered with Elpenhaler®db (Rolenium®) versus the innovative one (Seretide Diskus®)
  Other Names: Rolenium; Seretide

SUMMARY:
The aim of this study is to establish the therapeutic equivalence between the test (Fluticasone/Salmeterol administered with Elpenhaler®db, Rolenium®) and the reference formulation (Seretide®, administered with Diskus®), both containing 250/50μg of the Fluticasone/Salmeterol combination.

In case of inhaled products, it is not possible to follow the classic scheme, based on similarity of plasma concentration-time behavior of parent drug in assessing bioequivalence.

DETAILED DESCRIPTION:
A pharmacodynamic study was designed in order to assess the therapeutic equivalence of the new formulation of Fluticasone/Salmeterol with the innovative one. The test and reference Fluticasone/Salmeterol formulations will be compared in terms of their bronchodilator effects in lung function. Forced Expiratory Volume in 1 second (FEV1) will be the primary efficacy measure and will be measured in such a way that a similar time-dependent increase in pulmonary function can be demonstrated for both Fluticasone/Salmeterol formulations in patients with asthma. In terms of safety comparison, repeated measurements of adverse events, vital signs, heart rate, blood hematology and biochemistry as well as ECG changes will enable the establishment of the similar safety profile of the test and reference Fluticasone/Salmeterol combinations.

The study will be conducted in a randomized, double-blind, double-dummy, placebo-controlled, 3x3 crossover fashion.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years,
* diagnosis of asthma of 6 months,
* FEV1 ≥ 50% and ≤ 80% predicted, reversibility of at least 12%,
* stable asthma for at least 4 weeks,
* inhaled steroids (ICS) at a stable dose within the previous 30 days,
* PIF 30 - 90 lt/min and
* informed consent.

Exclusion Criteria:

* history of other pulmonary disease, asthma exacerbation or respiratory infection within the previous 4 weeks,
* hospitalization for acute asthmatic symptoms requiring parenteral steroids or oral steroid dose increase within the previous 30 days,
* heavy smokers,
* change of asthma medication within the previous 4 weeks, seasonal asthma alone,
* history of severe heart disease,
* pregnancy or lactation,
* use of a β-blocker, of a NSAID or an antiallergic/antihistaminic medication within 2 weeks prior to screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
FEV1 | 8 days
  12-hour average FEV1

SECONDARY OUTCOMES:
Adverse Events | 8 days
  Number of Adverse Events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Katalin Gömöri, Principal Investigator — Számítógépes Adatszolgáltató és Kereskedelmi Kft.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: PMID: 17523742 DOI: 10.2165/00044011-200525010-00001 — https://pubmed.ncbi.nlm.nih.gov/17523742/